CLINICAL TRIAL: NCT01916486
Title: Complex Mental and Social Activities to Promote Cognitive Function in Older Adults With Chronic Stroke: A Randomized Controlled Trial
Brief Title: Vitality: Promoting Cognitive Function in Older Adults With Chronic Stroke
Acronym: Vitality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-00715
Record Dates: First submitted 2013-07-23; First posted 2013-08-05 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Chronic Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise; Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise training (Experimental): Twice-weekly for the 6-month duration.
  Interventions: Behavioral: Exercise training
- Complex mental and social activities (Experimental): Twice-weekly for the 6-month duration.
  Interventions: Behavioral: Complex mental and social activities
- Control: stretching and relaxation program (Active Comparator): Twice-weekly for the 6-month duration.
  Interventions: Behavioral: Control: stretching and relaxation program

INTERVENTIONS:
Behavioral: Exercise training — The EX Program will provide objective progression in the guided exercises of each participant.
  Other Names: EX Program
  Arms: Exercise training
Behavioral: Complex mental and social activities — The Cog-Plus Program will engage participants in activities promoting cognitive function and socialization.
  Other Names: Cog-Plus Program
  Arms: Complex mental and social activities
Behavioral: Control: stretching and relaxation program — The CON Program consist of stretches, deep breathing and relaxation techniques, general posture education, and general core control exercises in the sitting position.
  Other Names: CON Program
  Arms: Control: stretching and relaxation program

SUMMARY:
The investigators will conduct a randomized controlled trial study to provide preliminary evidence of efficacy of exercise training or a complex mental and social activities program for improving cognitive function in older adults with chronic stroke, compared with a stretch and relaxation program.

DETAILED DESCRIPTION:
A total of 119 adults diagnosed with chronic stroke will be randomized to either a 6-month twice-weekly exercise program, complex mental and social activities program, or stretch and relaxation program. After 6 months of intervention, they will be followed for an additional 6 months. There will be four measurement sessions: baseline, 3 months, 6 months (end of intervention period); and 12 months.

ELIGIBILITY:
The study will specifically recruit individuals who had an ischemic or hemorrhagic stroke and have probable mild cognitive impairment.

In addition, individuals must meet the following inclusion criteria:

1. Aged 55 years or over;
2. Have a history of a single stroke of at least one year prior to study enrolment;
3. Mini-Mental State Examination (MMSE) (5) score of ≥ 20 at screening, including a perfect score on the 3-step command to ensure intact comprehension and ability to follow instructions;
4. Have subjective cognitive complaints;
5. Community-dwelling;
6. Lives in Metro Vancouver;
7. Able to comply with scheduled visits, treatment plan, and other trial procedures;
8. Must be able to read, write, and speak English in which psychometric tests are provided with acceptable visual and auditory acuity;
9. Stable on a fixed dose of cognitive medications (e.g., donepezil, galantamine, rivastigmine, memantine, etc.) that is not expected to change during the 12-month study period, or, if they are not on any of these medications, they are not expected to start them during the 12-month study period;
10. Able to walk for a minimum of six metres with rest intervals with or without assistive devices;
11. Have an activity tolerance of 60 minutes with rest intervals;
12. Not currently participating in any regular therapy or progressive exercise; and
13. Provide a personally signed and dated informed consent document indicating that the individual (or a legally acceptable representative) has been informed of all pertinent aspects of the trial. In addition, an assent form will be provided at baseline and again at regular intervals.

Exclusion Criteria:

1. Diagnosed with dementia of any type;
2. Diagnosed with another type of neurodegenerative or neurological condition (ie. Parkinson's disease) that affects cognitive function and mobility;
3. At high risk for cardiac complications during exercise and/or unable to self-regulate activity or to understand recommended activity level (i.e., Class C of the American Heart Risk Stratification Criteria);
4. Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility, as determined by his/her family physician;
5. Taking medications that may negatively affect cognitive function, such as anticholinergics, including agents with pronounced anticholinergic properties (e.g., amitriptyline), major tranquilizers (typical and atypical antipsychotics), and anticonvulsants (e.g., gabapentin, valproic acid, etc.); or
6. Have aphasia as judged by an inability to communicate by phone.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2019-08 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognitive function as measured by the Alzheimer's Disease Assessment Scale Cognitive Subscale Plus (ADAS-Plus) at 6 months | Baseline and 6 months
  ADAS-Cog 13 + additional measures of executive functions. For ADAS-Cog 13, higher scores indicate greater impairment.

SECONDARY OUTCOMES:
Change from baseline in executive functions as measured by the Stroop Test. | Baseline, 3 months (for subset of cognitive outcomes), 6 months, and 12 months
Change from baseline in executive functions as measured by the Tower of London Test. | Baseline, 3 months (for subset of cognitive outcomes), 6 months, and 12 months
Change from baseline in processing speed and executive functions as measured by the Trail Making Tests (Parts A & B). | Baseline, 3 months (for subset of cognitive outcomes), 6 months, and 12 months
Change from baseline in category fluency. | Baseline, 3 months (for subset of cognitive outcomes), 6 months, and 12 months
Change from baseline in memory and executive functions as measured by the verbal digits forward and backward tests. | Baseline, 3 months (for subset of cognitive outcomes), 6 months, and 12 months
Change from baseline in instrumental activities of daily living as measured by the Instrumental Activities of Daily Living Scale. | Baseline, 3 months, 6 months, and 12 months
  Higher scores indicate better performance.
Change from baseline in fatigue as measured by the Fatigue Severity Scale. | Baseline, 3 months, 6 months, and 12 months
  Higher scores indicate greater fatigue.
Change from baseline in physical activity level as measured by the Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS). | Baseline, 3 months, 6 months, and 12 months
  Acquired on a monthly basis. Higher scores indicate greater activity.
Change from baseline in community mobility as measured by the Life-space Assessment (LSA). | Baseline, 3 months, 6 months, and 12 months
  Higher scores indicate greater community mobility.
Change from baseline in leisure activity as measured by the Shortened Nottingham Leisure Scale. | Baseline, 3 months, 6 months, and 12 months
  Acquired on a monthly basis. Higher scores indicate greater leisure activity.
Change from baseline in general balance and mobility as measured by the Short Physical Performance Battery. | Baseline, 3 months, 6 months, and 12 months
Change from baseline in functional capacity as measured by the 6 Minute Walk Test. | Baseline, 3 months, 6 months, and 12 months
Change from baseline in general balance and mobility as measured the Timed Up-and-Go Test. | Baseline, 3 months, 6 months, and 12 months
Change from baseline in quadriceps strength. | Baseline, 3 months, 6 months, and 12 months
Change from baseline in grip strength. | Baseline, 3 months, 6 months, and 12 months
Change from baseline in mood as measured by the Center for Epidemiologic Studies Depression Scale. | Baseline, 3 months, 6 months, and 12 months
  Higher scores indicate greater impairment in mood.
Change from baseline in quality of life as measured by the European Quality of Life-5 Dimensions (EQ-5D). | Baseline, 3 months, 6 months, and 12 months
  Acquired on a monthly basis.
Change from baseline in quality of life as measured by European Quality of Life-5 Dimensions Visual Analog Scale (EQ-5D VAS). | Baseline, 3 months, 6 months, and 12 months
  Acquired on a monthly basis.
Change from Baseline in Cognitive Function as Measured by the Alzheimer's Disease Assessment Scale Cognitive Subscale Plus (ADAS-Cog Plus) at 12 months | Baseline, 3 months, 6 months, and 12 months
  ADAS-Cog 13 + additional measures of executive functions. For ADAS-Cog Plus, higher scores indicate greater impairment.
Change from Baseline in sleep quality as measured by the Pittsburgh Sleep Index. | Baseline, 3 months, 6 months, and 12 months
Change from Baseline in sleep quality as measured by the Motion Watch 8. | Baseline, 3 months, 6 months, and 12 months
Change from Baseline in lipid profile. | Baseline and 6 months
Change from Baseline in insulin sensitivity. | Baseline and 6 months
Health care resource usage. | Baseline, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janice J Eng, PhD, PT, Principal Investigator — University of British Columbia; Teresa Liu-Ambrose, PhD, PT, Principal Investigator — University of British Columbia; Peter Hall, PhD, Principal Investigator — University of Waterloo; Charlie Goldsmith, PhD, Principal Investigator — Simon Fraser University; Jennifer Davis, PhD, Principal Investigator — University of British Columbia; Laura Middleton, PhD, Principal Investigator — University of Waterloo; Ging-Yuek Robin Hsiung, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Liu-Ambrose T, Falck RS, Dao E, Best JR, Davis JC, Bennett K, Hall PA, Hsiung GR, Middleton LE, Goldsmith CH, Graf P, Eng JJ. Effect of Exercise Training or Complex Mental and Social Activities on Cognitive Function in Adults With Chronic Stroke: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2236510. doi: 10.1001/jamanetworkopen.2022.36510. PMID 36227593
- [Derived] Falck RS, Best JR, Davis JC, Eng JJ, Middleton LE, Hall PA, Liu-Ambrose T. Sleep and cognitive function in chronic stroke: a comparative cross-sectional study. Sleep. 2019 May 1;42(5):zsz040. doi: 10.1093/sleep/zsz040. PMID 30805652
- [Derived] Best JR, Eng JJ, Davis JC, Hsiung R, Hall PA, Middleton LE, Graf P, Goldsmith CH, Liu-Ambrose T. Study protocol for Vitality: a proof-of-concept randomised controlled trial of exercise training or complex mental and social activities to promote cognition in adults with chronic stroke. BMJ Open. 2018 Mar 17;8(3):e021490. doi: 10.1136/bmjopen-2018-021490. PMID 29550783